CLINICAL TRIAL: NCT06517615
Title: The Effect of Home Visit Supported Nursing Education Program on Some Parameters in Elderly People Living Alone at Home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Zeynep Arabacı, Public Health Nursing Dr., Kastamonu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KastamonuUniversity
Record Dates: First submitted 2024-04-29; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Old Age; Debility; Loneliness; Healthy Lifestyle
Keywords: elderly; home visit; nursing
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: The study was planned as a quasi-experimental research.
Masking Description: as a quasi-experimental research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial (Experimental): Home Visit Supported Nursing Training Program
  Interventions: Behavioral: Home Visit Supported Nursing Training Program
- control (No Intervention): standart care

INTERVENTIONS:
Behavioral: Home Visit Supported Nursing Training Program — Individualized Nurse Education Program with Home Visit Support (• Walking and exercise programs, Disease self-management training for those with chronic diseases, techniques and practices that facilitate medication compliance, vital sign monitoring, • • • Nutrition charts and follow-ups, food characteristics information and weight tracking, cooking activities in the kitchen,• Helping to create family and friend systems, creating neighbor communication mechanisms
  Arms: trial

SUMMARY:
It is aimed to develop healthy lifestyle behaviors of elderly people living alone at home, reduce their loneliness levels and increase their social support capacity.The research was planned as a quasi-experimental research. The research population consists of elderly people living alone at home who are registered to the Elderly and Home Care Unit of a Municipality of a province.

DETAILED DESCRIPTION:
When elderly people want to live in their own homes, an important issue arises: loneliness. Loneliness is a common problem among older adults and has become increasingly common in recent years. Loneliness not only affects psychological well-being, but also negatively affects physical health, increasing the likelihood of illness and death.When people live longer, they are more likely to experience health problems such as physical weakness, cognitive decline, and chronic diseases. Weakness among older people creates a state of vulnerability that increases the risk of adverse health outcomes, leading to reduced daily activities and the need for long-term care.This study aims to develop healthy lifestyle behaviors, reduce loneliness levels and increase social support capacity of elderly people living alone at home.The research was planned as a quasi-experimental research. The research population consists of elderly people living alone at home who are registered to the Elderly and Home Care Unit of a Municipality of a province. Elderly people who are registered to a home care unit, live alone, and are over the age of 65 and agree to work will be included in the research. Individuals under the age of 65 and those with mental disabilities will be excluded from the study. The independent variable of the research is; The status of receiving a home visit supported nurse care program was determined as the dependent variable of the study: Healthy Lifestyle Behaviors Scale II score, loneliness scale score, social support scale score.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older
* receiving home care services
* agreeing to participate in the study
* be literate

Exclusion Criteria:

* Individuals under the age of 65
* be mentally retarded
* not volunteering

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-12-29 (Estimated); Study Completion 2024-12-29 (Estimated)

PRIMARY OUTCOMES:
Healthy Lifestyle Behaviors Scale II score increase | 8 week
  Healthy Lifestyle Behaviors Scale II score
UCLA Loneliness Scale Short Form-6 point decrease | 8 week
  UCLA Loneliness Scale Short Form-6 point
Multidimensional Perceived Social Support Scale score increase | 8 week
  Multidimensional Perceived Social Support Scale score

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep ARABACI, Dr, Principal Investigator — zarabaci@kastamonu.edu.tr
Locations (2):
- Turkey (Türkiye) (2):
  - Kastamonu Üniversity, Kastamonu
  - Zeynep ARABACI, Kastamonu

IPD SHARING:
Plan to Share IPD: No